CLINICAL TRIAL: NCT06924528
Title: The Effects Of Toy In Chıldren Durıng Inhaler Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Ayse Boke, Principal Investigator, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BakırköySadiKonuk-aboke-01
Record Dates: First submitted 2025-04-05; First posted 2025-04-11 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Lower Respiratory Tract Disease; Respiratory Disease
Keywords: children; inhalation therapy; toy; anxiety; emotional state
MeSH Terms: conditions — Respiration Disorders; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The intervention group received the mask application on the toy. The control group did not receive the mask application on the toy.
Who Masked: Participant
Masking Description: Seventy-two participants included in the study were divided into two groups: intervention and control. The assignment of participants to the intervention and control groups was done randomly by someone not involved in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The control group (No Intervention): 5 minutes before starting the inhaler treatment, the child's anxiety level should be determined, and the child's emotional state should be evaluated by two observers.
  After washing hands, the aerosol medication ordered by the physician should be applied using a nebulizer mask.
  In the 5th minute after the inhaler treatment begins, the child's anxiety level should be determined, and the child's emotional state should be evaluated by two observers.
  5 minutes after the inhaler treatment ends, the child's anxiety level should be determined, and the child's emotional state should be evaluated by two observers.
- The intervention group (Experimental): 5 minutes before starting the inhaler treatment, the child's anxiety level should be determined, and the child's emotional state should be evaluated by two observers.
  After washing hands, the aerosol medication ordered by the physician should be applied using a nebulizer mask.
  The child is introduced to the plush toy of Kral Şakir, a character they recognize from cartoons. After explaining that King Şakir also needs help to recover, the nebulizer mask is applied to the toy, and saline solution is added to the mask's reservoir. Then, the treatment is started together with the child.
  In the 5th minute after the inhaler treatment begins, the child's anxiety level should be determined, and the child's emotional state should be evaluated by two observers.
  5 minutes after the inhaler treatment ends, the child's anxiety level should be determined, and the child's emotional state should be evaluated by two observers.
  Interventions: Other: using toy during inhaler treatment

INTERVENTIONS:
Other: using toy during inhaler treatment — The mask application on the toy will be performed only during the first inhaler treatment that the children receive in the emergency department.
  Other Names: using toy
  Arms: The intervention group

SUMMARY:
The purpose of the study is to investigate the effect of using a toy that children like during inhaler treatment on children's anxiety and emotional state. In the study, an inhaler treatment will be applied to children with a mask placed on a toy that they like. The purpose of this intervention is to reduce the child's anxiety and increase their emotional adjustment by improving adherence to the treatment.

DETAILED DESCRIPTION:
Respiratory diseases are commonly seen during childhood. Today, inhaler medication is frequently used in the treatment of lower respiratory tract diseases. Inhalation therapy is the process of delivering liquid medication in aerosol form directly to the respiratory tract and lungs using devices called nebulizers. Compared to other treatment methods, the direct delivery of medication to the lungs, the rapid onset of effect, and fewer systemic side effects make inhalation therapy the preferred method for treating children. In treatments administered through inhalation, if the inhalation is being applied for the first time, the child may experience fear and anxiety due to not knowing the procedure. After the nurse explains how the procedure is done, they should use distraction techniques to relax the child and support the effective continuation of the inhalation treatment. Distraction techniques are simple and inexpensive methods, and studies have proven their positive effect on children. This study is designed to investigate the effect of using a toy during inhaler treatment on children's anxiety and emotional state.

ELIGIBILITY:
Inclusion Criteria:

* The child being between the ages of 4 and 6,
* The child being scheduled to receive their first inhaler treatment after admission to the unit,
* No IV or IM interventions being performed before the inhaler treatment,
* The child and parents being willing to participate in the study,
* No mental or neurological disabilities present in the child or parent,
* The child not having any life-threatening illnesses,
* The child having an oxygen saturation of 95% or higher,
* The child's body temperature not exceeding 37.5 degrees Celsius,
* The child's cognitive level and motor development being appropriate for their age,
* The child being able to count up to 10,
* The parent being literate,
* No visual or auditory problems present in the child or parent

Exclusion Criteria:

* The child's general condition (tachycardia, fever, vomiting, etc.) and orientation (disorientation, lethargy, etc.) significantly deteriorating after the inhaler treatment begins,
* The parent or child wanting to withdraw from the study at any stage of the research.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2024-11-02 (Actual); Primary Completion 2025-03-26 (Actual); Study Completion 2025-04-05 (Actual)

PRIMARY OUTCOMES:
children's anxiety meter state | five months
  To measure state anxiety, children are asked to mark how they feel "right now." To measure trait anxiety, another copy of the scale is presented, and they are asked to mark how they "usually feel at home." Examples of being at home are provided to the children, like "think about when you were playing outside with a friend" and "think about sitting quietly watching TV." Before completing the scale, children were screened for their ability to rank order by size. They were asked to count to 10, and then answer, "Which is bigger, 7 or 4?" Children were also asked to identify the smallest of a series of four stacking cups. Children unable to complete these tasks successfully or who did not understand the instructions did not complete the scale.

SECONDARY OUTCOMES:
Children's Emotional Manifestation Scale | five months
  In the scale, emotional indicators are evaluated based on five parameters. These parameters are: facial expression, voice, activity, interaction, and cooperation level. Each of these five parameters is scored on a scale from 1 to 5, with the lowest possible score being "5" and the highest possible score being "25."
  In the first category, facial expression, the child's facial expressions observed by the researcher are scored on 5 items.
  Secondly, in the vocalization category, the child's tearfulness is evaluated through 5 sub-items.
  Thirdly, in the movement category, scoring is done based on the child's body language, using 5 sub-items.
  Fourthly, in the interaction category, the child's verbal and non-verbal communication is evaluated through 5 sub-items.
  Finally, in the cooperation category, the child's active or passive participation is observed and scored based on 5 sub-items.

CONTACTS AND LOCATIONS:
Locations (1):
- Bakirkoy Dr Sadi Konuk Researching and Training Hospital, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No